CLINICAL TRIAL: NCT04608643
Title: Correlation Between Inflammatory Markers and Complete Blood Film Indices (White Blood Cells and Platelets ) in Severely Malnourished Children
Brief Title: Inflammatory Markers and Cbc Indices in Severely Malnourished Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Meret Michael Fahmy, doctor, Assiut University
Other Study IDs: infection in malnutrition
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Response
Keywords: inflammatory markers in severly malnourished children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC _inflammatory markers _ platelet function test — CBC , Erythrocte sedimentation rate (ESR) ,CRP, platlet functions tests ( adhesions, 'aggregations ristocetin).

SUMMARY:
The main objectives of this study were to correlate between inflammatory markers and cbc indices in severly malnourished children and to determine whether children with SAM can mount an acute phase reactant response namely CRP and to evaluate the usefulness of quantitative CRP as a predictor of severe infections in children with SAM.

And to correlate between inflammatory markers and CBC indices (mainly white blood cells and platelets in those children .

DETAILED DESCRIPTION:
Malnutrition remains one of the most common causes of morbidity and mortality among children throughout the world.

Malnutrition is a pathological state resulting from a relative or absolute deficiency or excess of one or more essential nutrients it may be clinically manifested or detected by biochemical ,anthropometric measurements In 2009, the World Health Organization (WHO) estimated that 20 million children under 5 years suffered from severe acute malnutrition (SAM) worldwide, which is associated to more than half of their deaths each year in developing countries.

Severe acute malnutrition is defined by a very low weight for height ( below -3z scores of the median WHO growth standards ,by visible severe wasting or by presence of nutritional edema It diminishes immune function and prevents the host from mounting an adequate protective response to infectious agents. In turn, infections alter nutrient status and can create a deficiency state. Thus, malnutrition and infection often act synergistically to increase morbidity and mortality, particularly among infants and children The usual signs of infection are absent or nonspecific in children with acute severe malnutrition (SAM), Furthermore, laboratory diagnostic capacity is often limited in regions with the highest burdens of malnutrition.

Malnourished patients maintain the capacity to release inflammatory markers such as CRP & Interleukin-6 which can be considered favorable for combating infections.

Malnourished patients maintain the capacity to release inflammatory markers such as CRP which can be considered favorable for combating infections.

(CRP) as a diagnostic tool of infection in children by the fact that SAM, particularly edematous malnutrition, can be associated with reduced levels of acute phase proteins.

Malnutrition results in various changes in the body including changes in haematologic profile of the body. White cell changes seen in protein energy malnutrition varies and such changes have been attributed to various factors.

These include the synergist relationship which protein energy malnutrition has with infections and thymic atrophy seen in children with PEM also platlet count and function affected in SAM Various authors correlate blood platelet activation with infections and concluded that Platelet destruction occurs in infection and hypercoagulable state . Moreover, blood platelet has immunological functions and participate in the interaction between pathogens and host defenses . Other studies revealed that some platelets functions (ADP and collagen - induced platelets aggregations) have been decreased in protein energy malnutrition .

ELIGIBILITY:
Inclusion Criteria:

- All children aged 6 months up to 5 years who were admitted with the diagnosis of SAM .

The diagnosis of SAM was made using the recent WHO criteria measuring weight for length/height and mid-upper arm circumference (MUAC) and the presence of bilateral pitting oedema and severe wasting. Two forms of SAM exist in children: nonoedematous malnutrition, also known as marasmus, characterized by severe wasting and currently defined by weight for length/height z score < -3 of the WHO growth standard, or MUAC <11.5 cm; and edematious malnutrition defined by bilateral pitting edema also known as Kwashiorkor.10 The term marasmic kwashiorkor, has been used to describe children with both wasting and edema.

Exclusion Criteria:

* 1. Children below 6 months or above 5 years 2. Children with mild and moderate malnutrition, 3. Children with malnutrition secondary to serious underlying conditions including

  * Congenital anomalies, inborn errors of metabolism, malignancies, inherited autosomal disorders like cystic fibrosis, chronic diarrhial diseases like coeliac disease,
  * Congenital cardiac diseases, chronic kidney disease were excluded from the study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patients who are included with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
correlate between inflammatory markers and cbc indices in severly malnourished children | baseline
  to determine whether children with SAM can mount an acute phase reactant response namely CRP and to evaluate the usefulness of quantitative CRP as a predictor of severe infections in children with SAM.
  And to correlate between inflammatory markers and CBC indices (mainly WBCS and platelets in those children .

REFERENCES:
- [Background] Calder PC, Jackson AA. Undernutrition, infection and immune function. Nutr Res Rev. 2000 Jun;13(1):3-29. doi: 10.1079/095442200108728981. PMID 19087431
- [Background] Chisti MJ, Tebruegge M, La Vincente S, Graham SM, Duke T. Pneumonia in severely malnourished children in developing countries - mortality risk, aetiology and validity of WHO clinical signs: a systematic review. Trop Med Int Health. 2009 Oct;14(10):1173-89. doi: 10.1111/j.1365-3156.2009.02364.x. PMID 19772545
- [Background] Page AL, de Rekeneire N, Sayadi S, Aberrane S, Janssens AC, Rieux C, Djibo A, Manuguerra JC, Ducou-le-Pointe H, Grais RF, Schaefer M, Guerin PJ, Baron E. Infections in children admitted with complicated severe acute malnutrition in Niger. PLoS One. 2013 Jul 17;8(7):e68699. doi: 10.1371/journal.pone.0068699. Print 2013. PMID 23874731
- [Background] Delgado AF, Okay TS, Leone C, Nichols B, Del Negro GM, Vaz FA. Hospital malnutrition and inflammatory response in critically ill children and adolescents admitted to a tertiary intensive care unit. Clinics (Sao Paulo). 2008 Jun;63(3):357-62. doi: 10.1590/s1807-59322008000300012. PMID 18568246
- [Background] Jahoor F, Badaloo A, Reid M, Forrester T. Protein metabolism in severe childhood malnutrition. Ann Trop Paediatr. 2008 Jun;28(2):87-101. doi: 10.1179/146532808X302107. PMID 18510818
- [Background] Speth C, Loffler J, Krappmann S, Lass-Florl C, Rambach G. Platelets as immune cells in infectious diseases. Future Microbiol. 2013 Nov;8(11):1431-51. doi: 10.2217/fmb.13.104. PMID 24199802
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19087431/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=Pneumonia+in+severely+malnourished+children+in+developing+countries
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23874731/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/18568246/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/18510818/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/24199802/